CLINICAL TRIAL: NCT00686829
Title: Vicriviroc (SCH 417690) Treatment Protocol in HIV-Infected Subjects: A Rollover Study for ACTG Protocol A5211
Brief Title: Vicriviroc (SCH 417690) Treatment Protocol in Human Immunodeficiency Virus (HIV)-Infected Participants: A Rollover Study for ACTG Protocol A5211 (P04100)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04100; MK-7690-027 (Other: Merck Protocol Number)
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: HIV; HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — vicriviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VCV 30 mg (Experimental): Participants take VCV 30 mg once daily.
  Interventions: Drug: Vicriviroc maleate

INTERVENTIONS:
Drug: Vicriviroc maleate — VCV 30 mg tablet once daily by mouth.
  Other Names: SCH 417690

SUMMARY:
The purpose of this study is to provide open-label vicriviroc (VCV) to human immunodeficiency virus (HIV) treatment-experienced participants who successfully completed 48 weeks of treatment on Acquired Immunodeficiency Syndrome (AIDS) Clinical Trial Group (ACTG) protocol A5211 (or who responded favorably to treatment but discontinued participation due to viral tropism shifts), and participants who screened for ACTG A5211 and met all inclusion/exclusion criteria, but were unable to enroll due to protocol closure.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of ACTG Protocol A5211, or favorable response in A5211 but discontinued due to tropism shift, or screened for A5211 and met inclusion/exclusion criteria but unable to enroll due to protocol closure.
* Participants must also be on a ritonavir-containing antiretroviral regimen at entry, and have acceptable hematologic and laboratory parameters.
* Female participants of reproductive potential must agree to use 2 reliable methods of contraception, including a barrier method, and must have a negative urine pregnancy test prior to dosing.

Exclusion Criteria:

* History of seizure or drug use that increases risk of seizure, current use of CYP3A4 inducers, prior history of malignancy, active drug or alcohol use or dependence that would interfere with study requirements
* Female participants who are breast-feeding, pregnant, or plan to become pregnant
* Participation in a clinical trial with another investigational drug.
* Participants with serious illness requiring systemic therapy and/or hospitalization must not begin VCV (if not already on VCV) until participant completes therapy or is clinically stable on therapy for at least 14 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2005-06-30 (Actual); Primary Completion 2010-10-21 (Actual); Study Completion 2010-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Wilkin TJ, Su Z, Krambrink A, Long J, Greaves W, Gross R, Hughes MD, Flexner C, Skolnik PR, Coakley E, Godfrey C, Hirsch M, Kuritzkes DR, Gulick RM. Three-year safety and efficacy of vicriviroc, a CCR5 antagonist, in HIV-1-infected treatment-experienced patients. J Acquir Immune Defic Syndr. 2010 Aug;54(5):470-6. doi: 10.1097/qai.0b013e3181e2cba0. PMID 20672447
- [Result] Yeh TM, Evans SR, Gulick RM, Clifford DB. Vicriviroc and peripheral neuropathy: results from AIDS Clinical Trials Group 5211. HIV Clin Trials. 2010 Jan-Feb;11(1):51-8. doi: 10.1310/hct1101-51. PMID 20400411
- [Result] Tsibris AM, Paredes R, Chadburn A, Su Z, Henrich TJ, Krambrink A, Hughes MD, Aberg JA, Currier JS, Tashima K, Godfrey C, Greaves W, Flexner C, Skolnik PR, Wilkin TJ, Gulick RM, Kuritzkes DR. Lymphoma diagnosis and plasma Epstein-Barr virus load during vicriviroc therapy: results of the AIDS Clinical Trials Group A5211. Clin Infect Dis. 2009 Mar 1;48(5):642-9. doi: 10.1086/597007. PMID 19191652

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with human immunodeficiency virus (HIV) infection enrolled in AIDS Clinical Trial Group (ACTG) study A5211 (NCT00082498) and (1) completed the 48-week phase, or (2) had detectable alpha-chemokine receptor 4 (CXCR4)-tropic virus but maintained a virologic response and no drop in cluster of differentiation 4 (CD4)/CD8 count from baseline, or (3) met all inclusion/exclusion criteria but were unable to enroll in ACTG A5211 due to protocol closure prior to their randomization and dosing.
Groups:
- VCV 30 mg: Participants took VCV 30 mg once daily.
Period: Overall Study
Arm/Group | VCV 30 mg
Started (Number of participants who were previously enrolled in study ACTG A5211 who received ≥1 dose of VCV in P04100.) | 79
Completed | 0
Not Completed | 79
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 6
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 14
Not completed — Protocol Violation | 3
Not completed — Sponsor discontinued VCV | 47

BASELINE CHARACTERISTICS:
Arm/Group | VCV 30 mg
Number analyzed (Participants) | 79
Age, Continuous [Mean (Full Range); unit: Years] | 49 [30 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 60
  More than one race | 4
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With ≥1 Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product, biologic (at any dose), or medical device, which does not necessarily have a causal relationship with the treatment.
Time Frame: Up to discontinuation of commercial VCV availability (up to approximately 5.5 years)
Population: All treated participants are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | VCV 30 mg
Number analyzed (Participants) | 79
Percentage of Participants | 91

2. Primary Outcome: Percentage of Participants Discontinuing Study Therapy Due to AEs
Description: as for outcome 1
Time Frame: Up to discontinuation of commercial VCV availability (up to approximately 5.5 years)
Population: All treated participants are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | VCV 30 mg
Number analyzed (Participants) | 79
Percentage of Participants | 6

3. Primary Outcome: Percentage of Participants With ≥1 Serious Adverse Events (SAEs)
Description: An SAE is any adverse occurrence that results in death; is life-threatening; results in a persistent disability; requires in-patient hospitalization or prolongs hospitalization; or is a congenital anomaly/birth defect.
Time Frame: Up to discontinuation of commercial VCV availability (up to approximately 5.5 years)
Population: All treated participants are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | VCV 30 mg
Number analyzed (Participants) | 79
Percentage of Participants | 48

4. Primary Outcome: Percentage of Participants With HIV Ribonucleic Acid (RNA) <50 Copies/mL
Description: The percentage of participants with HIV RNA <50 copies/mL at each time point is reported. For this measure, "month" was defined as each 28-day period on study treatment. The Roche Amplicor® HIV-1 monitor test was used to quantify HIV RNA.
Time Frame: Every 12 months up to 60 months
Population: All treated participants with HIV RNA data available are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | VCV 30 mg
Number analyzed (Participants) | 79
Percentage of Participants
  Month 12: number analyzed (Participants) | 60
  Month 12 | 52
  Month 24: number analyzed (Participants) | 53
  Month 24 | 64
  Month 36: number analyzed (Participants) | 49
  Month 36 | 80
  Month 48: number analyzed (Participants) | 44
  Month 48 | 89
  Month 60: number analyzed (Participants) | 20
  Month 60 | 80

5. Primary Outcome: Percentage of Participants With HIV RNA >50 to <400 Copies/mL
Description: The percentage of participants with HIV RNA >50 to <400 copies/mL at each time point is reported. For this measure, "month" was defined as each 28-day period on study treatment. The Roche Amplicor® HIV-1 monitor test was used to quantify HIV RNA.
Time Frame: Every 12 months up to 60 months
Population: All treated participants with HIV RNA data available are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | VCV 30 mg
Number analyzed (Participants) | 79
Percentage of Participants
  Month 12: number analyzed (Participants) | 60
  Month 12 | 13
  Month 24: number analyzed (Participants) | 53
  Month 24 | 11
  Month 36: number analyzed (Participants) | 49
  Month 36 | 12
  Month 48: number analyzed (Participants) | 44
  Month 48 | 2
  Month 60: number analyzed (Participants) | 20
  Month 60 | 15

6. Primary Outcome: Percentage of Participants With HIV RNA ≥400 Copies/mL
Description: The percentage of participants with HIV RNA ≥400 copies/mL at each time point is reported. For this measure, "month" was defined as each 28-day period on study treatment. The Roche Amplicor® HIV-1 monitor test was used to quantify HIV RNA.
Time Frame: Every 12 months up to 60 months
Population: All treated participants with HIV RNA data available are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | VCV 30 mg
Number analyzed (Participants) | 79
Percentage of Participants
  Month 12: number analyzed (Participants) | 60
  Month 12 | 35
  Month 24: number analyzed (Participants) | 53
  Month 24 | 25
  Month 36: number analyzed (Participants) | 49
  Month 36 | 8
  Month 48: number analyzed (Participants) | 44
  Month 48 | 9
  Month 60: number analyzed (Participants) | 20
  Month 60 | 5

7. Primary Outcome: Number of Participants With Coreceptor Tropism Shifts From Baseline
Description: The number of participants with non reportable (NR) tropism, CCR5 (R5) tropism, or dual/mixed CCR5/CXCR4 (DM/X4) tropism at baseline, who had NR, R5, or DM/X4 tropism at the time of virologic failure (VF) is reported. The definition of VF is an increase in HIV RNA level >0.5 log10 copies/mL compared to the baseline HIV RNA level.
Time Frame: Baseline (Week 48 of ACTG study A5211) and time of VF in P4100, assessed up to approximately 5.5 years
Population: All treated participants with baseline and VF tropism data available are included.
Measure: Number; unit: Participants
Arm/Group | VCV 30 mg
Number analyzed (Participants) | 79
Participants
  NR Baseline to NR VF: number analyzed (Participants) | 60
  NR Baseline to NR VF | 45
  NR at Baseline to R5 VF: number analyzed (Participants) | 60
  NR at Baseline to R5 VF | 10
  NR Baseline to DM/X4 VF: number analyzed (Participants) | 60
  NR Baseline to DM/X4 VF | 5
  R5 baseline to R5 VF: number analyzed (Participants) | 15
  R5 baseline to R5 VF | 11
  R5 baseline to NR VF: number analyzed (Participants) | 15
  R5 baseline to NR VF | 3
  R5 baseline to DM/X4 VF: number analyzed (Participants) | 15
  R5 baseline to DM/X4 VF | 1
  DM/X4 baseline to DM/X4 VF: number analyzed (Participants) | 4
  DM/X4 baseline to DM/X4 VF | 3
  DM/X4 baseline to R5 VF: number analyzed (Participants) | 4
  DM/X4 baseline to R5 VF | 1

8. Primary Outcome: Mean Change From Baseline in CD4/CD8 Cell Counts
Description: The mean change from baseline in CD4/CD8 counts throughout P4100 until the time of VF is reported. "Month" was defined as each 28-day period on study treatment. A fluorescent-activated cell sorter (FACS) analysis was used to quantify CD4/CD8 lymphocytes. The definition of VF is an increase in HIV RNA level >0.5 log10 copies/mL compared to the baseline HIV RNA level.
Time Frame: Baseline (Week 48 of ACTG study A5211) and up to time of VF in P4100, assessed up to approximately 5.5 years
Population: All treated participants with baseline and on-treatment CD4/CD8 data available are included.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | VCV 30 mg
Number analyzed (Participants) | 79
cells/mm^3
  Month 2: number analyzed (Participants) | 54
  Month 2 | -16.26 (103.83)
  Month 4: number analyzed (Participants) | 64
  Month 4 | -17.70 (84.87)
  Month 6: number analyzed (Participants) | 61
  Month 6 | 9.30 (95.38)
  Month 8: number analyzed (Participants) | 59
  Month 8 | -0.20 (115.96)
  Month 10: number analyzed (Participants) | 58
  Month 10 | 12.59 (97.84)
  Month 12: number analyzed (Participants) | 58
  Month 12 | -13.81 (124.09)
  Month 14: number analyzed (Participants) | 61
  Month 14 | 18.56 (106.18)
  Month 16: number analyzed (Participants) | 57
  Month 16 | 21.63 (130.33)
  Month 18: number analyzed (Participants) | 58
  Month 18 | 2.82 (108.52)
  Month 20: number analyzed (Participants) | 54
  Month 20 | 19.71 (125.34)
  Month 22: number analyzed (Participants) | 51
  Month 22 | 24.19 (94.37)
  Month 24: number analyzed (Participants) | 47
  Month 24 | 32.04 (121.45)
  Month 26: number analyzed (Participants) | 49
  Month 26 | 34.36 (128.99)
  Month 28: number analyzed (Participants) | 49
  Month 28 | 36.10 (120.75)
  Month 30: number analyzed (Participants) | 49
  Month 30 | 38.10 (113.80)
  Month 32: number analyzed (Participants) | 46
  Month 32 | 47.59 (137.15)
  Month 34: number analyzed (Participants) | 46
  Month 34 | 61.93 (109.71)
  Month 36: number analyzed (Participants) | 46
  Month 36 | 43.63 (136.85)
  Month 38: number analyzed (Participants) | 43
  Month 38 | 90.81 (140.11)
  Month 40: number analyzed (Participants) | 45
  Month 40 | 75.53 (142.90)
  Month 42: number analyzed (Participants) | 40
  Month 42 | 104.65 (187.14)
  Month 44: number analyzed (Participants) | 44
  Month 44 | 91.61 (181.71)
  Month 46: number analyzed (Participants) | 42
  Month 46 | 91.19 (165.33)
  Month 48: number analyzed (Participants) | 42
  Month 48 | 93.93 (174.36)
  Month 50: number analyzed (Participants) | 41
  Month 50 | 128.12 (189.94)
  Month 52: number analyzed (Participants) | 44
  Month 52 | 107.41 (170.97)
  Month 54: number analyzed (Participants) | 34
  Month 54 | 136.00 (211.98)
  Month 56: number analyzed (Participants) | 31
  Month 56 | 129.87 (196.80)
  Month 58: number analyzed (Participants) | 21
  Month 58 | 188.81 (152.93)
  Month 60: number analyzed (Participants) | 20
  Month 60 | 122.60 (191.32)
  Month 62: number analyzed (Participants) | 13
  Month 62 | 132.54 (118.87)
  Month 64: number analyzed (Participants) | 10
  Month 64 | 147.50 (197.12)
  Month 66: number analyzed (Participants) | 2
  Month 66 | 283.50 (2.12)
  Month 68: number analyzed (Participants) | 2
  Month 68 | 300.00 (50.91)

9. Primary Outcome: Number of Participants With Reduced Susceptibility to VCV
Description: The total number of participants with viruses having phenotypic resistance to VCV is reported. Viruses exhibiting both maximum percent inhibition (MPI) plateau values of <85% and relative MPI (R-MPI) values of <0.9 (based on the PhenoSense HIV entry assay) were considered to have phenotypic resistance to VCV.
Time Frame: Up to time of VF in P4100, assessed up to approximately 5.5 years
Population: All treated participants are included.
Measure: Number; unit: Participants
Arm/Group | VCV 30 mg
Number analyzed (Participants) | 79
Participants | 7

10. Primary Outcome: Number of Participants With AIDS-defining Events (ADEs)
Description: The number of participants with ADEs is reported. An ADE is an SAE that is expected in the course of disease and not considered related to study intervention. The sponsor identified events that met ADE criteria based on the 1993 Centers for Disease Control (CDC) Revised Classification System.
Time Frame: Up to discontinuation of commercial VCV availability (up to approximately 5.5 years)
Population: All treated participants are included.
Measure: Number; unit: Participants
Arm/Group | VCV 30 mg
Number analyzed (Participants) | 79
Participants
  Plasmablastic Lymphoma | 1
  Kaposi's Sarcoma | 1

11. Primary Outcome: Number of Participants With New Infections
Description: The number of participants with new infections is reported.
Time Frame: Up to discontinuation of commercial VCV availability (up to approximately 5.5 years)
Population: All treated participants are included.
Measure: Number; unit: Participants
Arm/Group | VCV 30 mg
Number analyzed (Participants) | 79
Participants
  Herpes simplex virus infection | 6
  Upper respiratory tract infection | 39

ADVERSE EVENTS:
Time Frame: Up to approximately 5.5 years
Description: All treated participants are included.
Arm/Group | VCV 30 mg
All-Cause Mortality (participants affected / at risk) | 3/79
Serious Adverse Events (participants affected / at risk) | 38/79
Other Adverse Events (participants affected / at risk) | 70/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VCV 30 mg (N=79)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1)
ARRHYTHMIA (Cardiac disorders) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (2)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 3 (3)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1)
PERICARDITIS (Cardiac disorders) | 1 (1)
SICK SINUS SYNDROME (Cardiac disorders) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1)
EYELID PTOSIS (Eye disorders) | 1 (1)
GLAUCOMA (Eye disorders) | 1 (1)
OPTIC ISCHAEMIC NEUROPATHY (Eye disorders) | 1 (1)
RETINAL VEIN OCCLUSION (Eye disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 2 (2)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (2)
OESOPHAGEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
PARAESTHESIA ORAL (Gastrointestinal disorders) | 1 (1)
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
SWOLLEN TONGUE (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 2 (3)
ASTHENIA (General disorders) | 1 (1)
CHEST PAIN (General disorders) | 3 (3)
CHILLS (General disorders) | 1 (1)
PYREXIA (General disorders) | 3 (3)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1)
ALLERGY TO VACCINE (Immune system disorders) | 1 (1)
ANOGENITAL WARTS (Infections and infestations) | 2 (2)
ARTHRITIS BACTERIAL (Infections and infestations) | 1 (1)
BACTERAEMIA (Infections and infestations) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (2)
CELLULITIS (Infections and infestations) | 3 (3)
ENDOCARDITIS BACTERIAL (Infections and infestations) | 1 (1)
MENINGITIS COCCIDIOIDES (Infections and infestations) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 5 (5)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
STAPHYLOCOCCAL ABSCESS (Infections and infestations) | 1 (1)
VIRAL PERICARDITIS (Infections and infestations) | 1 (1)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1)
BLOOD AMYLASE INCREASED (Investigations) | 3 (3)
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 1 (2)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1)
LIPASE INCREASED (Investigations) | 2 (2)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 2 (2)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1)
AXILLARY MASS (Musculoskeletal and connective tissue disorders) | 1 (1)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
ANAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1)
MUSCLE CONTRACTIONS INVOLUNTARY (Nervous system disorders) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 1 (1)
ALCOHOL ABUSE (Psychiatric disorders) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5 (7)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 (1)
CARDIAC PACEMAKER REVISION (Surgical and medical procedures) | 1 (1)
COLOSTOMY (Surgical and medical procedures) | 1 (1)
HIP ARTHROPLASTY (Surgical and medical procedures) | 1 (1)
HYSTERECTOMY (Surgical and medical procedures) | 1 (1)
LAMINAPLASTY (Surgical and medical procedures) | 1 (1)
LARGE INTESTINE ANASTOMOSIS (Surgical and medical procedures) | 1 (1)
OESOPHAGOGASTRIC FUNDOPLASTY (Surgical and medical procedures) | 1 (1)
SIGMOIDECTOMY (Surgical and medical procedures) | 1 (1)
EMBOLISM ARTERIAL (Vascular disorders) | 1 (1)
HAEMATOMA (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VCV 30 mg (N=79)
EAR CONGESTION (Ear and labyrinth disorders) | 4 (4)
EYE PAIN (Eye disorders) | 4 (5)
EYE PRURITUS (Eye disorders) | 4 (4)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 9 (15)
ABDOMINAL PAIN (Gastrointestinal disorders) | 11 (18)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 7 (10)
CONSTIPATION (Gastrointestinal disorders) | 9 (13)
DIARRHOEA (Gastrointestinal disorders) | 26 (44)
DYSPEPSIA (Gastrointestinal disorders) | 5 (6)
FLATULENCE (Gastrointestinal disorders) | 5 (5)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 9 (10)
HAEMATOCHEZIA (Gastrointestinal disorders) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 28 (43)
TOOTHACHE (Gastrointestinal disorders) | 5 (8)
VOMITING (Gastrointestinal disorders) | 11 (17)
CHEST DISCOMFORT (General disorders) | 4 (4)
CHEST PAIN (General disorders) | 5 (9)
CHILLS (General disorders) | 8 (11)
FATIGUE (General disorders) | 29 (44)
OEDEMA PERIPHERAL (General disorders) | 8 (12)
PAIN (General disorders) | 6 (7)
PYREXIA (General disorders) | 18 (27)
BRONCHITIS (Infections and infestations) | 11 (12)
CELLULITIS (Infections and infestations) | 4 (6)
HERPES SIMPLEX (Infections and infestations) | 4 (4)
HERPES ZOSTER (Infections and infestations) | 7 (10)
NASOPHARYNGITIS (Infections and infestations) | 6 (6)
OTITIS MEDIA (Infections and infestations) | 4 (4)
PNEUMONIA (Infections and infestations) | 8 (9)
SINUSITIS (Infections and infestations) | 15 (24)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 18 (28)
URINARY TRACT INFECTION (Infections and infestations) | 5 (5)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 5 (8)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (5)
BLOOD AMYLASE INCREASED (Investigations) | 6 (9)
BLOOD GLUCOSE INCREASED (Investigations) | 6 (10)
WEIGHT DECREASED (Investigations) | 6 (6)
DECREASED APPETITE (Metabolism and nutrition disorders) | 6 (9)
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 9 (9)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 4 (5)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 4 (4)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 14 (36)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 13 (18)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 7 (8)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 4 (4)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 12 (17)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 4 (5)
MYALGIA (Musculoskeletal and connective tissue disorders) | 10 (12)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 6 (7)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 25 (53)
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (6)
DIZZINESS (Nervous system disorders) | 16 (24)
HEADACHE (Nervous system disorders) | 20 (28)
HYPOAESTHESIA (Nervous system disorders) | 14 (21)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 5 (7)
PARAESTHESIA (Nervous system disorders) | 11 (11)
ANXIETY (Psychiatric disorders) | 9 (10)
DEPRESSION (Psychiatric disorders) | 13 (15)
INSOMNIA (Psychiatric disorders) | 13 (13)
MICTURITION URGENCY (Renal and urinary disorders) | 4 (5)
NEPHROLITHIASIS (Renal and urinary disorders) | 4 (6)
POLLAKIURIA (Renal and urinary disorders) | 5 (7)
COUGH (Respiratory, thoracic and mediastinal disorders) | 23 (42)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 11 (20)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 5 (7)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 14 (29)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 10 (13)
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 5 (5)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 10 (13)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 6 (9)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 5 (7)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 4 (6)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 5 (7)
PRURITUS (Skin and subcutaneous tissue disorders) | 4 (6)
RASH (Skin and subcutaneous tissue disorders) | 9 (11)
SINUS OPERATION (Surgical and medical procedures) | 5 (5)
HYPERTENSION (Vascular disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation with regard to (1) proprietary information that is protected by the provisions contained in paragraph B below, (2) the accuracy of the information contained in the publication, and (3) to ensure that the presentation is fairly balanced and in compliance with FDA regulations.